CLINICAL TRIAL: NCT05782985
Title: Expression Pattern of Heterogeneous Nuclear Ribonucleoprotein H1 (HNRNPH1) and K (HNRNPK) Genes in Myeloproliferative Neoplasms
Brief Title: Expression Pattern of HNRNPH1 and HNRNPK Genes in MPNs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed Mohamed Kamal Elminshawy, Assistant Lecturer, Assiut University
Other Study IDs: HNRNPH1 & HNRNPK in MPNs
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Myeloproliferative Neoplasms (MPNs)
Keywords: heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1); heterogeneous nuclear ribonucleoprotein K (HNRNPK); Myeloproliferative Neoplasms (MPNs)
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myeloproliferative neoplasms Cases: The myeloproliferative neoplasms Cases will be tested for expression of heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) and K (HNRNPK) genes
  Interventions: Diagnostic Test: Reverse transcription-quantitative polymerase chain reaction (RT-qPCR)
- Controls: Healthy controls will be tested for expression of heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) and K (HNRNPK) genes
  Interventions: Diagnostic Test: Reverse transcription-quantitative polymerase chain reaction (RT-qPCR)

INTERVENTIONS:
Diagnostic Test: Reverse transcription-quantitative polymerase chain reaction (RT-qPCR) — Blood samples from the myeloproliferative neoplasms cases and the controls will be tested with Reverse transcription-quantitative polymerase chain reaction (RT-qPCR) for expression of heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) and K (HNRNPK) genes.

SUMMARY:
The aim of the study is to evaluate the expression pattern of heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) and K (HNRNPK) genes in Myeloproliferative neoplasms as a possible indicator of disease progression and as a potential therapeutic target

DETAILED DESCRIPTION:
Self-renewing Hematopoietic pluripotent stem cells can develop into either myeloid or lymphoid lineages. A diverse range of diseases known as myeloproliferative neoplasms (MPNs) develop due to the aberrant proliferation of one or more terminal myeloid cell lines in the peripheral circulation. MPNs come in four traditional forms: chronic myeloid leukaemia (CML), polycythaemia vera (PV), essential thrombocythemia (ET), and primary myelofibrosis (PMF). Chronic neutrophilic leukaemia (CNL), chronic eosinophilic leukaemia (CEL), and MPN unclassifiable, were also included in the WHO classification. While PV, ET, and PMF are BCR-ABL1 negative, CML is BCR-ABL1 positive.

In eukaryotic cell's nucleus, many ribonucleoproteins (RNPs) assemble on to recently produced transcripts. The heterogeneous nuclear ribonucleoproteins (hnRNPs) are one type of RNPs. Some hnRNPs are now known to play a role in the development of human hematologic malignancies. Disease research is becoming more interested in how hnRNPs control gene expression. Numerous cancers exhibit changed hnRNPs expression levels, which raises the possibility that they play a part in carcinogenesis.

For instance, leukaemia cells showed downregulation of Heterogeneous nuclear ribonucleoprotein K (HNRNPK). In vivo myeloproliferative neoplasm tumour growth was accelerated by HNRNPK knockdown. On the other hand, A study suggests that HNRNPK overexpression could accelerate CML development and thus a possible indicator of CML progression and a potential therapeutic target might be HNRNPK.

Moreover, one of the earliest RNA-binding proteins (RBPs) to be identified, Heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) contributes to RNA stabilization, RNA editing, and RNA modification. Previous research has demonstrated that high levels of HNRNPH1 expression leads to carcinogenesis by both upregulating the expression of oncogenes and downregulating the expression of tumour suppressor genes such P53, Ron, and BCL-X.

The investigators performed the study with the aim to study the expression level of heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) and K (HNRNPK) genes and their proteins in MPNs and to investigate the association of HNRNPH1 and HNRNPK with molecular diagnostic tests of MPNs.

ELIGIBILITY:
Inclusion Criteria:

The study will be carried out on patients newly diagnosed with one of the myeloproliferative neoplasms based on WHO Criteria for diagnosis of MPNs whether males or females and of any age.

Exclusion Criteria:

* Other malignancies.
* Patients on chemotherapy or radiotherapy.
* Autoimmune diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed myeloproliferative neoplasms patients
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Expression of Heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) and Heterogeneous nuclear ribonucleoprotein K (HNRNPK) genes in myeloproliferative neoplasms (MPNs) | two years
  Expression levels of Heterogeneous nuclear ribonucleoprotein H1 (HNRNPH1) and Heterogeneous nuclear ribonucleoprotein K (HNRNPK) genes for diagnosis of myeloproliferative neoplasms.

SECONDARY OUTCOMES:
Correlation between expression levels of HNRNPH1 and HNRNPK genes and molecular diagnostic tests for myeloproliferative neoplasms | Two years
  Correlation between expression levels of HNRNPH1 and HNRNPK genes and molecular diagnostic tests for myeloproliferative neoplasms as Philadelphia chromosome or JAK2 V617F or JAK2 exon 12 mutation or CALR or MPL mutation according to the case

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Elminshawy, MD, Mac, Principal Investigator — Assiut University
Locations (1):
- Assiut University Department of Clinical Pathology, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Tefferi A, Thiele J, Vardiman JW. The 2008 World Health Organization classification system for myeloproliferative neoplasms: order out of chaos. Cancer. 2009 Sep 1;115(17):3842-7. doi: 10.1002/cncr.24440. PMID 19472396
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] Gallardo M, Lee HJ, Zhang X, Bueso-Ramos C, Pageon LR, McArthur M, Multani A, Nazha A, Manshouri T, Parker-Thornburg J, Rapado I, Quintas-Cardama A, Kornblau SM, Martinez-Lopez J, Post SM. hnRNP K Is a Haploinsufficient Tumor Suppressor that Regulates Proliferation and Differentiation Programs in Hematologic Malignancies. Cancer Cell. 2015 Oct 12;28(4):486-499. doi: 10.1016/j.ccell.2015.09.001. Epub 2015 Sep 24. PMID 26412324
- [Background] Dreyfuss G, Matunis MJ, Pinol-Roma S, Burd CG. hnRNP proteins and the biogenesis of mRNA. Annu Rev Biochem. 1993;62:289-321. doi: 10.1146/annurev.bi.62.070193.001445. No abstract available. PMID 8352591
- [Background] Du Q, Wang L, Zhu H, Zhang S, Xu L, Zheng W, Liu X. The role of heterogeneous nuclear ribonucleoprotein K in the progression of chronic myeloid leukemia. Med Oncol. 2010 Sep;27(3):673-9. doi: 10.1007/s12032-009-9267-z. Epub 2009 Aug 4. PMID 19653139
- [Background] Han SP, Tang YH, Smith R. Functional diversity of the hnRNPs: past, present and perspectives. Biochem J. 2010 Sep 15;430(3):379-92. doi: 10.1042/BJ20100396. PMID 20795951
- [Background] Garneau D, Revil T, Fisette JF, Chabot B. Heterogeneous nuclear ribonucleoprotein F/H proteins modulate the alternative splicing of the apoptotic mediator Bcl-x. J Biol Chem. 2005 Jun 17;280(24):22641-50. doi: 10.1074/jbc.M501070200. Epub 2005 Apr 18. PMID 15837790
- [Background] Decorsiere A, Cayrel A, Vagner S, Millevoi S. Essential role for the interaction between hnRNP H/F and a G quadruplex in maintaining p53 pre-mRNA 3'-end processing and function during DNA damage. Genes Dev. 2011 Feb 1;25(3):220-5. doi: 10.1101/gad.607011. PMID 21289067
- [Background] Braun S, Enculescu M, Setty ST, Cortes-Lopez M, de Almeida BP, Sutandy FXR, Schulz L, Busch A, Seiler M, Ebersberger S, Barbosa-Morais NL, Legewie S, Konig J, Zarnack K. Decoding a cancer-relevant splicing decision in the RON proto-oncogene using high-throughput mutagenesis. Nat Commun. 2018 Aug 17;9(1):3315. doi: 10.1038/s41467-018-05748-7. PMID 30120239
- [Background] Panelli D, Lorusso FP, Papa F, Panelli P, Stella A, Caputi M, Sardanelli AM, Papa S. The mechanism of alternative splicing of the X-linked NDUFB11 gene of the respiratory chain complex I, impact of rotenone treatment in neuroblastoma cells. Biochim Biophys Acta. 2013 Feb;1829(2):211-8. doi: 10.1016/j.bbagrm.2012.12.001. Epub 2012 Dec 12. PMID 23246602